CLINICAL TRIAL: NCT00856011
Title: Posterior Interosseous Nerve Pathology May Provide Novel Insights Into Both Predisposition and Potential Vascular Basis for the Development of Carpal Tunnel Syndrome in Diabetic Patients.
Brief Title: Nerve Morphology in Diabetic Patients
Status: Completed | Type: Observational
Sponsor: Skane University Hospital (Other)
Responsible Party: Niels Thomsen, MD
Other Study IDs: LU 508-03 (2003)
Record Dates: First submitted 2009-03-04; First posted 2009-03-05 (Estimated); Last update posted 2009-03-05 (Estimated); Status verified 2009-03

CONDITIONS: Peripheral Neuropathy; Carpal Tunnel Syndrome; Entrapment Neuropathies; Diabetes Complications
MeSH Terms: conditions — Peripheral Nervous System Diseases; Carpal Tunnel Syndrome; Nerve Compression Syndromes; Diabetes Complications

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Biopsies of the posterior interosseous nerve
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Diabetic patients with carpal tunnel syndrome
- 2: Non-diabetic patients with carpal tunnel syndrome

SUMMARY:
The underlying basis of carpal tunnel syndrome and the basis of its increased incidence in diabetes are unknown. The aim of this study was to quantified pathology in an uncompressed nerve (posterior interosseous nerve in the forearm between diabetic and non-diabetic patients with CTS.

ELIGIBILITY:
Inclusion Criteria

* Diagnosis of carpal tunnel syndrome based in clinical history and symptoms
* Confirmed by nerve conduction studies

Exclusion Criteria

* Other focal nerve entrapments
* Cervical radiculopathy
* Inflammatory joint disease
* Renal failure
* Thyroid disorders
* Previous wrist fracture
* Long-term exposure to vibrating tools
* Age under 18

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred to a specialized hand clinic
Sampling Method: Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2003-12; Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Nerve morphology (Fascicular area, myelinated nerve fiber density, endoneurial capillary density and subperineurial space

CONTACTS AND LOCATIONS:
Locations (1):
- Dept. of Hand Surgery, Malmo University Hospital, Malmo, Sweden